CLINICAL TRIAL: NCT00555672
Title: A Phase I Study Of Sunitinib Malate In Combination With Cisplatin And 5-Fluorouracil In Patients With Advanced Gastric Cancer
Brief Title: Study Of Sunitinib In Combination With Cisplatin And 5-Fluorouracil In Patients With Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181128
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Results first posted 2011-01-05 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil; Cisplatin; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: 5-fluorouracil; Drug: cisplatin; Drug: sunitinib malate

INTERVENTIONS:
Drug: 5-fluorouracil — 5- fluorouracil is given as 4000 mg/m^2 total dose over 96 hr continuous infusion of a 21 day chemotherapy cycle. Each 21 day cycle is repeated until progression of disease or unacceptable toxicity is observed.
Drug: cisplatin — Cisplatin is given 80 mg/m^2 through a vein on day 1 every 21 days. Each 21 day cycle is repeated until progression of disease or unacceptable toxicity is observed.
Drug: sunitinib malate — sunitinib is given orally 37.5mg /day for 14 days followed by 7 days of drug free period. Each 21 day cycle is repeated until progression of disease or unacceptable toxicity is observed.

SUMMARY:
The purpose of this study is to determine the safe and tolerable dose of sunitinib when given together with cisplatin and 5-fluorouracil in patients with advanced gastric cancer who have not received prior chemotherapy for their advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of stomach cancer
* advanced stomach cancer stage IV
* adequate blood chemistry, blood counts and kidney function
* willing to participate to study requirements and to sign an informed consent document

Exclusion Criteria:

* prior chemotherapy for stomach cancer in its advanced stage
* excessive toxicities related to prior therapies
* pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Spain (3):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181128&StudyName=Study%20Of%20Sunitinib%20In%20Combination%20With%20Cisplatin%20And%205-Fluorouracil%20In%20Patients%20With%20Advanced%20Gastric%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib (25 mg) in Combination With Cisplatin and 5-FU: Sunitinib: 25 milligram (mg) oral capsule daily for 2 weeks (Day 1 to 14) followed by 1 week (Day 15 to 21) off treatment. Cisplatin: 80 mg per meter squared (mg/m^2) intravenous on Day 1 of each 21-day cycle. 5-Fluorouracil (5-FU): 4000 mg/m^2 continuous infusion for 96 hours starting Day 1 and ending Day 5 of each 21-day cycle.
- Sunitinib (37.5 mg) in Combination With Cisplatin and 5-FU: Sunitinib: 37.5 mg oral capsule daily for 2 weeks (Day 1 to 14) followed by 1 week (Day 15 to 21) off treatment. Cisplatin: 80 mg per meter squared (mg/m^2) on Day 1 of each 21-day cycle. 5-Fluorouracil (5-FU): 4000 mg/m^2 continuous infusion for 96 hours starting Day 1 and ending Day 5 of each 21-day cycle.
Period: Overall Study
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU | Sunitinib (37.5 mg) in Combination With Cisplatin and 5-FU
Started | 24 | 10
Completed | 0 | 0
Not Completed | 24 | 10
Not completed — Death | 0 | 2
Not completed — Adverse Event | 8 | 2
Not completed — Objective progression or relapse | 11 | 5
Not completed — Other | 3 | 1
Not completed — Participant refused | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU | Sunitinib (37.5 mg) in Combination With Cisplatin and 5-FU | Total
Number analyzed (Participants) | 24 | 10 | 34
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (12.0) | 56.4 (10.4) | 59.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 17 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First-cycle Dose Limiting Toxicities (DLTs)
Description: The incidence of DLTs assessed during the first cycle (21 days).
Time Frame: Cycle 1 (Baseline to Day 21)
Population: Safety: enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU | Sunitinib (37.5 mg) in Combination With Cisplatin and 5-FU
Number analyzed (Participants) | 24 | 10
Participants | 1 | 0

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 1 of Cycle 1 (2, 4, 6, 8, 10, and 24 hours post dose)
Population: Pharmacokinetic (PK): participants who received Sunitinib and had sufficient plasma concentration data for calculation of PK parameters; N=number of participants contributing to summary statistics. Cmax of Sunitinib, SU012662, and Total Drug (Sunitinib + SU012662) calculated for at least 6 individual participants treated at maximum tolerated dose.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU
Number analyzed (Participants) | 9
nanograms per milliliter (ng/mL)
  Sunitinib | 16.8 (8.19)
  SU012662 (metabolite of Sunitinib) | 2.24 (1.29)
  Total Drug (Sunitinib + SU012662) | 19.0 (9.35)

3. Secondary Outcome: Area Under the Curve From Time 0 to 24 Hours Postdose [AUC (0-24)]
Description: Area under the plasma concentration versus time curve from time 0 (pre-dose) to 24 hours postdose (0-24).
Time Frame: Day 1 of Cycle 1 (2, 4, 6, 8, 10, and 24 hours postdose)
Population: PK; N=the number of participants contributing to the summary statistics. AUC(0-24) of Sunitinib, SU012662, and Total Drug (Sunitinib + SU012662) calculated for at least 6 individual participants treated at the maximum tolerated dose (MTD; 25 mg Sunitinib).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU
Number analyzed (Participants) | 9
ng*h/mL
  Sunitinib | 249 (127)
  SU012662 (metabolite of Sunitinib) | 34.0 (19.5)
  Total Drug (Sunitinib + SU012662) | 283 (144)

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Tmax is the time to first occurrence of maximum observed plasma concentration (Cmax).
Time Frame: Day 1 of Cycle 1 (2, 4, 6, 8, 10, and 24 hours post dose)
Population: PK; N=the number of participants contributing to the summary statistics. Tmax of Sunitinib, SU012662, and Total Drug (Sunitinib + SU012662) calculated for at least 6 individual participants treated at the MTD (25 mg Sunitinib).
Measure: Median (Full Range); unit: hours
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU
Number analyzed (Participants) | 9
hours
  Sunitinib | 4.00 [2.00 to 24.0]
  SU012662 (metabolite of Sunitinib) | 4.00 [2.00 to 24.0]
  Total Drug (Sunitinib + SU012662) | 4.00 [2.00 to 24.0]

5. Secondary Outcome: Steady State Concentration (Css) of 5-Fluorouracil (5-FU)
Description: Steady state plasma concentration of 5-FU equals AUC(2-6) divided by 4, where AUC(2-6) is the area under the plasma concentration versus time curve from time 2 to 6 hours postdose (2-6).
Time Frame: Day 1 of Cycle 1 (2, 4, and 6 hours post infusion)
Population: PK; N=number of participants contributing to the summary statistics. Css calculated for at least 6 individual participants treated at the MTD (25 mg Sunitinib).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU
Number analyzed (Participants) | 6
ng/mL | 593 (433)

6. Secondary Outcome: Infusion Rate (Zero Order) (R0) of 5-FU
Description: Infusion rate of 5-FU equals total dose divided by infusion time.
Time Frame: Day 1 of Cycle 1 (2, 4, and 6 hours post infusion)
Population: PK; N= number of participants contributing to the summary statistics. R0 calculated for at least 6 individual participants treated at the MTD (25 mg Sunitinib).
Measure: Mean (Standard Deviation); unit: mg/hr
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU
Number analyzed (Participants) | 6
mg/hr | 68.2 (12.5)

7. Secondary Outcome: Clearance (CLss) of 5-FU
Description: Steady state total body clearance equals infusion rate (zero order) divided by steady state plasma concentration of 5-FU (R0/Css).
Time Frame: Day 1 of Cycle 1 (2, 4, and 6 hours post infusion)
Population: PK; N=the number of participants contributing to the summary statistics. CLss calculated for at least 6 individual participants treated at the MTD (25 mg Sunitinib).
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU
Number analyzed (Participants) | 6
Liters per hour | 161 (93.2)

8. Secondary Outcome: Area Under the Curve From Time 2 to 6 Hours Postdose [AUC (2-6)] of 5-FU
Description: Area under the plasma concentration versus time curve from time 2 to 6 hours postdose (2-6).
Time Frame: Day 1 of Cycle 1 (2, 4, and 6 hours post infusion)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU
Number analyzed (Participants) | 6
ng*h/mL | 2372 (1729)

9. Secondary Outcome: Number of Participants With Objective Response
Description: Number of participants with an objective response-based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR defined as the disappearance of all target lesions. PR defined as greater than or equal to (≥) 30 percent (%) decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline, Day 21 of every even-numbered cycle up to 15 Months
Population: Efficacy: all participants enrolled in the study who received at least 1 dose of study medication. N=number of participants with measurable disease at baseline.
Measure: Number; unit: Participants
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU | Sunitinib (37.5 mg) in Combination With Cisplatin and 5-FU
Number analyzed (Participants) | 23 | 10
Participants | 6 | 3
Statistical Analysis 1: Comparison: Sunitinib (25 mg) in Combination With Cisplatin and 5-FU vs Sunitinib (37.5 mg) in Combination With Cisplatin and 5-FU; Test type: Superiority or Other; Fisher Exact; Exact Method based on the F Distribution; Objective Response Rate (ORR) (percent) = 27.3, 95% CI 2-sided [13.3 to 45.5]

10. Secondary Outcome: Duration of Response (DR)
Description: Time from the first objective documentation of tumor response (confirmed or partial response) to first documented objective tumor progression or death due to any cause, whichever occurrs first. DR calculated as (Months) equals (the end date for DR minus first subsequent confirmed CR or PR plus 1) divided by 30.
Time Frame: Baseline up to Month 15
Population: Efficacy; N=number of participants with objective response.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU | Sunitinib (37.5 mg) in Combination With Cisplatin and 5-FU
Number analyzed (Participants) | 6 | 3
Months | 4.17 (2.28) | 4.13 (0.73)

11. Secondary Outcome: Progression-Free Survival (PFS)
Description: Median time (50%) from the first dose of study treatment to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first. PFS calculated as (Months) equals (first event date minus first dose date plus 1) divided by 30.
Time Frame: Baseline up to Month 15
Population: Efficacy
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU | Sunitinib (37.5 mg) in Combination With Cisplatin and 5-FU
Number analyzed (Participants) | 24 | 10
Months | 5.2 [3.8 to 7.6] | 6.2 [3.3 to 6.9]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU | Sunitinib (37.5 mg) in Combination With Cisplatin and 5-FU
Serious Adverse Events (participants affected / at risk) | 7/24 | 5/10
Other Adverse Events (participants affected / at risk) | 24/24 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU (N=24) | Sunitinib (37.5 mg) in Combination With Cisplatin and 5-FU (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Device occlusion (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 3
Pyrexia (General disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (25 mg) in Combination With Cisplatin and 5-FU (N=24) | Sunitinib (37.5 mg) in Combination With Cisplatin and 5-FU (N=10)
Anaemia (Blood and lymphatic system disorders) | 12 | 6
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 21 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 5
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 6 | 4
Aerophagia (Gastrointestinal disorders) | 2 | 0
Anal pruritus (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 9 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 14 | 4
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 13 | 9
Asthenia (General disorders) | 19 | 7
Chest pain (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 5
Medical device complication (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 19 | 8
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 2
Pain (General disorders) | 3 | 1
Pyrexia (General disorders) | 3 | 4
Jaundice (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 1 | 2
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 12 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 5 | 2
Dysgeusia (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Neurotoxicity (Nervous system disorders) | 4 | 0
Paraesthesia (Nervous system disorders) | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Renal artery thrombosis (Renal and urinary disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 1
Iliac artery thrombosis (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 2 | 0
Pallor (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.